CLINICAL TRIAL: NCT02163083
Title: Detection of Lymph Nodes by Means of Intraoperative Fluorescence Lymphography Using Indocyanine Green (ICG) During the Radical Robot-assisted Prostatectomy
Brief Title: Detection of Lymphnodes Using ICG During RARP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital Gronau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U1111-1157-6624; 2013-609-f-S (Other: ethical review committee)
Record Dates: First submitted 2014-06-10; First posted 2014-06-13 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lymphadenectomy using standard Methods (No Intervention): Lymphadenectomy will be performed as a standard procedure
- Lymphadenectomy using ICG (Experimental): A fluorescent dye (indocyanine green) will be ultrasound-controlled preoperatively injected in the prostate. During robot-assisted radical intervention by DaVinci ® robot the lymphadenectomy is performed using the fluorescence lymphography.
  Interventions: Procedure: ICG

INTERVENTIONS:
Procedure: ICG — Improvement of detection of positive lymphnodes
  Other Names: indocyanine green powder; Pulsion Medical Systems, München, Germany
  Arms: Lymphadenectomy using ICG

SUMMARY:
The purpose of this study is to investigate, whether the detection of lymph nodes by means of intraoperative fluorescence lymphography as part of lymphadenectomy in robot-assisted radical prostatectomy is higher than without the use of indocyanine green (ICG).

DETAILED DESCRIPTION:
ICG is a fluorescent dye that fluoresces green bound to proteins under illumination in the near-infrared range. Using this dye allows to visualize lymphatic nodes, by being injected into the tumor or directly surrounding tissue.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally limited prostate cancer;
* Intermediate or high risk tumor
* Recommended and planned prostatectomy;
* Completed and signed written consent;
* Voluntarily agreement to participate in this study
* Age of the study participants ≥ 18 years.

Exclusion Criteria:

* Allergic reaction to active ingredient (indocyanine green);
* Iodine allergy;
* Hyperthyroidism;
* High-grade renal impairment;
* High-grade hepatic insufficiency;
* Unwillingness to the storage and disclosure of pseudonymous disease and personal data
* psychiatric pre-existing conditions or other circumstances that make a cooperation by the patient in question

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The total number of detection rate of (positive) lymph nodes using ICG | during the surgery

SECONDARY OUTCOMES:
Measurements of the time, that takes to remove the lymph nodes | During the surgery

OTHER OUTCOMES:
Determine the anatomical location of the ICG-positive lymph node | During th surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jörn H. Witt, MD, Principal Investigator — St. Antonius Hospital Gronau
Locations (1):
- St. Antonius Hospital Gronau, Department for Urology, Pediatric Urology and Urologic Oncology, Gronau, Moellenweg 22, Germany

IPD SHARING:
Plan to Share IPD: No